CLINICAL TRIAL: NCT04081389
Title: Phase I Clinical Trial Assessing the Combination of Chemokine Modulation With Neoadjuvant Chemotherapy in Triple Negative Breast Cancer
Brief Title: Chemokine Modulation Therapy and Standard Chemotherapy Before Surgery for the Treatment of Early Stage Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 73718; NCI-2019-05299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 73718 (Other: Roswell Park Cancer Institute); UL1TR001412 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-09-09 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Early-Stage Breast Carcinoma; Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Celecoxib; Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes; Introns; Interferon alpha-2; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CKM weeks 1-3, doxorubicin, cyclophosphamide) (Experimental): Patients receive celecoxib PO BID, recombinant interferon alfa-2b IV over 20 minutes, and rintatolimod IV on days 1-3 of weeks 1-3, as well as paclitaxel IV over 1 hour once weekly on day 1. Treatment continues for a total of 12 weeks in the absence of disease progression or unacceptable toxicity. 1-3 weeks after last dose of paclitaxel, patients receive doxorubicin IV over 10 minutes and cyclophosphamide IV over 30 minutes. Treatment repeats every 2 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Celecoxib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Paclitaxel; Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod

INTERVENTIONS:
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Recombinant Interferon Alfa-2b — Given IV
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen

SUMMARY:
This phase I trial studies how well chemokine modulation therapy and standard chemotherapy given before surgery work in treating patients with early stage triple negative breast cancer. Chemokine modulation therapy, including celecoxib, recombinant interferon alfa-2b, and rintatolimod, may stimulate the immune system and stop tumor cells from growing. Drugs used in standard chemotherapy, such as paclitaxel, doxorubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemokine modulation therapy together with standard chemotherapy may work better than giving either therapy alone in treating patients with triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the safety and tolerability profile of the combination of rintatolimod celecoxib +/- interferon alpha-2b, when given as CKM along with chemotherapy in the neoadjuvant setting in early stage triple negative breast cancer.

II To identify the appropriate dose level of CKM and paclitaxel for future clinical exploration.

SECONDARY OBJECTIVES:

II. • Evaluate the effect of neoadjuvant CKM + paclitaxel on pathological response and breast MRI response in early stage triple negative breast cancer patients.

III. • Evaluate the overall and recurrence-free survival in early stage triple negative breast cancer patients that received neoadjuvant CKM + paclitaxel.

EXPLORATORY OBJECTIVES:

I• To evaluate longitudinal changes of blood biomarkers such as peripheral T-cell subsets, myeloid derived suppressor cells (MDSC), expression of chemokine and other immune genes, circulating immune mediators and correlate them with the clinical course post surgery.

II• Comparison of response assessment criteria for a prospective analysis using RECIST 1.1. and irRECIST

* Evaluate changes in the intratumoral levels of biomarkers, such as, peripheral T-cell subsets, myeloid derived suppressor cells (MDSC), chemokines, and immune-regulatory factors (pre- vs post-CKM + paclitaxel treatment).

OUTLINE: This is a phase Ib, dose-escalation study of recombinant interferon alfa-2b.

Patients receive celecoxib orally (PO) twice daily (BID), recombinant interferon alfa-2b intravenously (IV) over 20 minutes (omitted in lowest dose level), and rintatolimod IV on days 1-3 of weeks 1-3, as well as paclitaxel IV over 1 hour once weekly on day 1. Treatment continues for a total of 12 weeks in the absence of disease progression or unacceptable toxicity. 1-3 weeks after last dose of paclitaxel, patients receive doxorubicin IV over 10 minutes and cyclophosphamide IV over 30 minutes. Treatment repeats every 2 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.

. After completion of study treatment, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed diagnosis of resectable triple negative breast cancer (ASCO/CAP guidelines will be used to define triple negative breast cancer)
* Must have measurable disease. Multi-centric disease is allowed. If patient has another lesion which is biopsied with ER/PR positive it will be Physician discretion for this eligibility criteria.
* Prior therapy: No prior cytotoxic regimens are allowed for this malignancy. Participants may not have had prior chemotherapy, other targeted anticancer therapies, or prior radiation therapy to the ipsilateral breast for this malignancy. Prior bis-phosphonate therapy is allowed
* Patient eligible for surgery as determined by patient's surgeon
* Patient must have a lesion that amendable to biopsy, unless inaccessible and with PI approval
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to swallow and retain oral medication
* Ability to undergo magnetic resonance imaging (MRI)
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and ALT (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 X institutional upper limit of normal (ULN)
* Creatinine < ULN OR creatinine clearance >= 50 mL/min per Cockcroft-Gault equation for patients with creatinine levels greater than ULN
* Left ventricular ejection fraction (LVEF) >= 55%; if LVEF is < 55% and patient is otherwise study-eligible, the principal investigator (PI) will discuss with cardiologist if patient is eligible to receive doxorubicin and participate in study
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Participants on this study will be counseled on and are willing to use adequate contraceptive methods

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment
* Patients with active autoimmune disease, requiring ongoing immunosuppressive therapy or history of transplantation
* Diagnosis of invasive carcinoma within the last 3 years
* Inflammatory breast cancer will be excluded from the study
* Participants who have metallic surgical implants that are not compatible with an MRI machine are not eligible
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Patients with known serious mood disorders. (Major depression is an exclusion. Other stable mood disorders on stable therapy for > 6 months may be allowed after consultation with PI)
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent
  * Patients with a New York Heart Association classification of III or IV
* History of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years
* Prior allergic reaction or hypersensitivity to nonsteroidal anti-inflammatory drugs (NSAIDs) or any drugs administered on protocol
* Any history of allergy to sulfonamides
* Any history of autoimmune hepatitis
* Grade 1 or higher neuropathy
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shipra Gandhi, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Interferon Alpha-2b at DL 1: Dose Level 1
  Celecoxib: 200 mg orally BID on days 1-3 of weeks 1-3.
  Interferon alpha-2b: None
  Rintatolimod: 200 mg intravenous on days 1-3 of weeks 1-3.
  Paclitaxel: 80 mg/m2 intravenous once weekly on day 1
- Arm 2: Interferon Alpha-2b at DL 2: Dose Level 2
  Celecoxib: 200 mg orally BID on days 1-3 of weeks 1-3.
  Interferon alpha-2b: 5 million units/m2 IV on days 1-3 of weeks 1-3.
  Rintatolimod: 200 mg intravenous on days 1-3 of weeks 1-3.
  Paclitaxel: 80 mg/m2 intravenous once weekly on day 1
- Arm 3: Interferon Alpha-2b at DL 3: Dose Level 3
  Celecoxib: 200 mg orally BID on days 1-3 of weeks 1-3.
  Interferon alpha-2b: 10 million units/m2 IV on days 1-3 of weeks 1-3.
  Rintatolimod: 200 mg intravenous on days 1-3 of weeks 1-3.
  Paclitaxel: 80 mg/m2 intravenous once weekly on day 1
- Arm 4: Interferon Alpha-2b at DL 4: Dose Level 4
  Celecoxib: 200 mg orally BID on days 1-3 of weeks 1-3.
  Interferon alpha-2b: 20 million units/m2 IV on days 1-3 of weeks 1-3.
  Rintatolimod: 200 mg intravenous on days 1-3 of weeks 1-3.
  Paclitaxel: 80 mg/m2 intravenous once weekly on day 1
Period: Overall Study
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
Started | 1 | 1 | 4 | 3
Completed | 1 | 1 | 3 | 3
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4 | Total
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (0) | 40.5 (0) | 45.7 (8.7) | 52.6 (4.6) | 47.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 3 | 9
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 3 | 3 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 4 | 3 | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Scale
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 0 | 1 | 4 | 3 | 8
    1 | 1 | 0 | 0 | 0 | 1
Overall American Joint Committee on Cancer (AJCC) Stage [Count of Participants; unit: Participants] — Increased stage corresponds to increased disease burden
  Stage 0 Stage I Stage II Stage III Stage IV
  Participants
    Stage I | 0 | 0 | 0 | 1 | 1
    Stage II | 1 | 0 | 2 | 0 | 3
    Stage III | 0 | 1 | 2 | 2 | 5
Laterality [Count of Participants; unit: Participants] — Side of cancer in breast.
  Participants
    Right Breast | 1 | 1 | 2 | 1 | 5
    Left Breast | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities
Description: Safety and toxicity will be assessed using the CTEP NCI Common Terminology Criteria for Adverse Events (CTCAE Version 5.0). The resulting dose limiting toxicity (DLT) information is used to identify the appropriate dose level of CKM and paclitaxel for future clinical exploration.
  The following events will be considered a DLT:
  * The event occurs within 3 weeks following 1st dose of combination CKM + paclitaxel therapy and subsequent enrollment for dose-escalation will only proceed after the 3-week period has been completed.
  * The toxicity has been determined by the investigator to be possibly, probably or definitely related to celecoxib, rintatolimod, interferon-α2b or paclitaxel.
  * Any death not clearly due to th
Time Frame: Within 21 days of treatment adminstration
Population: 1 patient was not DLT evaluable in DL3.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
Number analyzed (Participants) | 1 | 1 | 3 | 3
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Pathological Complete Response (pCR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI, where Complete Response (CR) corresponds to the disappearance of all target lesions.
Time Frame: Up to 4 week post-treatment (with a range of 7 to 11 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
Number analyzed (Participants) | 1 | 1 | 4 | 3
Participants | 0 | 1 | 2 | 2

3. Secondary Outcome: Residual Cancer Burden Index
Description: The calculated RCB index value is categorized as one of four RCB classes, RCB-0 to RCB-III where RCB-0 is best prognosis (no residual disease) to RCB-III a worst prognosis.
Time Frame: At 12 weeks post treatment initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
Number analyzed (Participants) | 1 | 1 | 4 | 3
Participants
  RCB-0 | 0 | 1 | 2 | 2
  RCB-I | 0 | 0 | 1 | 1
  RCB-II | 1 | 0 | 1 | 0

4. Secondary Outcome: Recurrence-free Survival (RFS)
Description: RFS is defined as local/regional invasive recurrence, invasive ipsilateral breast tumor recurrence, distant recurrence, inoperable (meaning no surgery because of progression), and/or death from breast cancer (per standard of care according to physician discretion) or any cause. RFS will be calculated from the time of treatment to event. The median RFS was estimated using standard Kaplan-Meier methods (where NR = not reached).
Time Frame: At 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
Number analyzed (Participants) | 1 | 1 | 4 | 3
months | 12.0 [NA to NA] — Unable to estimate the upper and lower bounds by the Kaplan-Meier method due to the number of observations (n=1). | NA [NA to NA] — No events observed, cannot estimate the median and corresponding bounds. | 11.4 [6.1 to 11.7] | 11.5 [11.4 to NA] — Unable to estimate the upper bound by the Kaplan-Meier method due to the limited number of events.

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined by death from breast cancer, non-breast cancer, unknown, or any other cause and will be calculated from the time of study entry to event. The median OS is estimated using standard Kaplan-Meier methods (where NR = not reached).
Time Frame: At 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
Number analyzed (Participants) | 1 | 1 | 4 | 3
months | 21.7 [NA to NA] — Unable to estimate the upper and lower bounds by the Kaplan-Meier method due to a sample size of n=1. | NA [NA to NA] — No events observed, cannot estimate the median and corresponding bounds. | NA [23.8 to NA] — Unable to estimate the upper bound by the Kaplan-Meier method due to the limited number of events. | NA [NA to NA] — No events observed, cannot estimate the median and corresponding bounds.

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 days after the final treatment administration (ranging from 7 to 11 weeks). All-cause mortality was monitored up to 3 years after treatment initiation.
Description: Grading scales found in the CTEP Version 5 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) will be utilized for AE reporting.
Arm/Group | Arm 1: Interferon Alpha-2b at DL 1 | Arm 2: Interferon Alpha-2b at DL 2 | Arm 3: Interferon Alpha-2b at DL 3 | Arm 4: Interferon Alpha-2b at DL 4
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/4 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Interferon Alpha-2b at DL 1 (N=1) | Arm 2: Interferon Alpha-2b at DL 2 (N=1) | Arm 3: Interferon Alpha-2b at DL 3 (N=4) | Arm 4: Interferon Alpha-2b at DL 4 (N=3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Interferon Alpha-2b at DL 1 (N=1) | Arm 2: Interferon Alpha-2b at DL 2 (N=1) | Arm 3: Interferon Alpha-2b at DL 3 (N=4) | Arm 4: Interferon Alpha-2b at DL 4 (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 4 (4) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (6) | 1 (1) | 2 (2) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (5) | 2 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (6) | 3 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (6) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (5) | 1 (1) | 3 (7) | 3 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (10) | 1 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 1 (2) | 4 (5) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04081389/Prot_SAP_000.pdf